CLINICAL TRIAL: NCT00925977
Title: Treatment Satisfaction of Insulin Glargine Plus Insulin Apidra Compared With NPH Insulin Plus Insulin Apidra in Recently Diagnosed Type 1 Diabetes Children and Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: rmc005275ctil
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Type 1
Keywords: treatment satisfaction; insulin Glargine; insulin Apidra; NPH insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- insulin Glargine + insulin Apidra (Active Comparator): insulin Glargine + insulin Apidra
  Interventions: Drug: insulin Glargine + Insulin Apidra
- Insulin NPH + Insulin Apidra (Active Comparator): 12 weeks treatment with Insulin NPH + Insulin Apidra
  Interventions: Drug: Insulin NPH + Insulin Apidra: Active Comparator

INTERVENTIONS:
Drug: insulin Glargine + Insulin Apidra — 12 wees treatment with Insulin Glargine + Insulin Apidra
  Arms: insulin Glargine + insulin Apidra
Drug: Insulin NPH + Insulin Apidra: Active Comparator — Insulin NPH + Insulin Apidra: Active Comparator
  Arms: Insulin NPH + Insulin Apidra

SUMMARY:
A randomized, crossover, open study in order to compare treatment satisfaction with insulin Glargine plus insulin Apidra Vs NPH insulin plus insulin Apidra in newly diagnosed children and adolescents with type 1 diabetes.

The study will include two consecutive periods: 2 weeks run in period and 24 weeks intervention period, divided into two separate treatment periods of 12 weeks. According to randomization, each patient will be treated consecutively with both treatment arms: 12 weeks with insulin Glargine and than 12 weeks with NPH insulin or 12 weeks with insulin NPH ad than 12 weeks with insulin Glargine. Patients will complete DTSQ (Diabetes Treatment Satisfaction Questionnaire) at months 0, 12 and 24 weeks, before and at the end of each study arm.

DETAILED DESCRIPTION:
A randomized, crossover, open study in order to compare treatment satisfaction with insulin Glargine plus insulin Apidra Vs NPH insulin plus insulin Apidra in newly diagnosed children and adolescents with type 1 diabetes.

134 Patients with new onset Diabetes type 1, diagnosed 12 months previously at maximum will be enrolled.

The study will include two consecutive periods: 2 weeks run in period and 24 weeks intervention period, divided into two separate treatment periods of 12 weeks. According to randomization, each patient will be treated consecutively with both treatment arms: 12 weeks with insulin Glargine and than 12 weeks with NPH insulin or 12 weeks with NPH insulin and than 12 weeks with insulin Glargine.

The study will consist of 4 clinical visits, taking place at -2, 0, 12 and 24 weeks. Height,weight,vital signs, HbA1c and insulin doses will be determined during the clinical visits.

Patients will complete DTSQ (Diabetes Treatment Satisfaction Questionnaire) at months 0, 12 and 24 weeks, before and at the end of each study arm.

The DTSQ questionnaires consists of DTSQ parents- for patients below the age of 13, and DTSQ teen for those above age 13.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes diagnosed less than 12 months prior to study entry
2. Age: 7-20 years old.
3. HbA1c>/=8.0
4. Signing inform consent form

Exclusion Criteria:

1. Any significant disease or conditions, including psychiatric disorders that in the opinion of the investigator are likely to effect his compliance or ability to complete the study.
2. Patients participating in other device or drug studies.
3. Any contraindication to insulin glargine and or insulin Apidra and or Insulin NPH according to SmPC.
4. Inability, of adolescent or parent, to understand/complete the Treatment satisfaction questionnaire.

Ages: 7 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Treatment satisfaction | patients will complete DTSQ at months 0,12 and 24

SECONDARY OUTCOMES:
HbA1c | value of Hba1C will be measured at screening visit and at the end of each study arm
4 and 7 points glucose profile | patients will complete a diary before all clinical visits
Insulin doses | Insulin doses will be determined at baseline visit and every visit after
Hypoglycemic events | patients will report in their diary every episode of hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Professor, Principal Investigator — Rabin Medical Center
Locations (4):
- Israel (4):
  - Soroka hospital, Bear Sheva
  - Rambam Hospital, Haifa
  - Health care unit- Jerusalem, Jerusalem
  - Schnider children medical center, Petah Tikva